CLINICAL TRIAL: NCT02673892
Title: The Impact of a Patient-Centered Discharge Summary (PODS) on Patient Experience and Health Outcomes Following Discharge: A Multicenter Randomized Controlled Trial
Brief Title: Patient Oriented Discharge Summary Impact Study
Acronym: PODS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recommendation of DMC - challenges recruiting, statistical considerations
Sponsor: University Health Network, Toronto (Other)
Collaborators: Baycrest (Other); Bruyère Health Research Institute. (Other); Thunder Bay Regional Health Sciences Centre (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15-9735-AE
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-04

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Pneumonia; Hip Fracture; Total Hip Replacement; Total Knee Replacement
Keywords: discharge; transitions; patient experience
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Pneumonia; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PODS intervention (Experimental): The PODS intervention is administered during the discharge process which includes discharge teaching. In the acute settings, discharge teaching is provided by a nurse navigator, resident physician, or other members of the care team. In the rehabilitation setting, discharge teaching is provided by a multi-disciplinary team. PODS is used as a useful add-on to the usual discharge teaching process. The PODS form used during the study will be a fillable pdf. Members of the healthcare team will fill it out electronically, then print it out and give the paper to the patient. After the discharge teaching is finished, patients take the completed PODS home with them as a post-discharge reference and guide.
  Interventions: Other: Patient Oriented Discharge Summary
- Usual Care (No Intervention): Patients randomized to this arm will receive usual discharge care. At UHN, this involves receiving a discharge summary with information pertaining to hospital course including investigations performed and medications used, as well as follow-up care suggested. It is intended to be, unlike PODS, a document for the primary care physician seeing the patient after discharge to refer to. As to discharge instructions provided for the patient, there is no standard procedure and sometimes follow-up instructions are included for the patient. Patient education may or may not be provided to the patient verbally by their nurse, resident, physician, or pharmacist. Moreover, follow-up with the primary care physician may be set up prior to or following discharge with the nurse navigator.

INTERVENTIONS:
Other: Patient Oriented Discharge Summary — The PODS provides a written template for providers to engage patients and caregivers when reviewing important discharge instructions on medications, activity and diet restrictions, follow-up appointments and worrisome symptoms warranting emergency care. The PODS also uses plain and simple wording, large fonts, pictograms, and includes white space for patients to take notes and provides the option for translation of major headings into the most common spoken languages. As this will be a pragmatic design, we may make modifications to the process involved in completing the PODS, such as using pre-filled disease-specific information, if system processes and providers involved deem it more usable and feasible.
  Arms: PODS intervention

SUMMARY:
Improving the patient experience has become a major focus of quality improvement efforts in Ontario and in health systems worldwide. However, our existing knowledge base is relatively under-developed, particularly in how patients experience care as they transition from one care setting to another and the relationship between patient experience and clinical outcomes. The Patient Oriented Discharge Summary (PODS) is a discharge instruction tool created by patients, caregivers, health-care providers and design experts. It provides a written template for providers to engage patients and caregivers when reviewing important instructions on medications, activity and diet restrictions, follow-up appointments and worrisome symptoms warranting emergency care following admission to hospital. The PODS also uses plain and simple wording, large fonts, pictograms, and includes white space for patients to take notes and provides the option for translation of major headings into the most common spoken languages. The PODS impact study will study the impact of using the PODS versus usual discharge instructions on patient experience and health outcomes in a provincial-wide randomized study across acute care and rehabilitation hospitals.

DETAILED DESCRIPTION:
Full Title: The impact of a patient-centered discharge summary (PODS) on patient experience and health outcomes following discharge: A multicenter randomized controlled trial.

Short Title: PODS Impact Study

Primary Objective: To evaluate the impact of a patient-centered discharge instruction tool on patient experience following hospital discharge.

Primary Outcome Measure: Patient experience within 72 hours following discharge from hospital. Count of negative responses (i.e., "No", or "Not at all" or "Partly") to 6 prespecified questions on patient experience of transition of care answered 72 hours following discharge from hospital, with the first 5 questions from the CIHI Patient Experiences Survey - In-Patient Care (CPES-IC). Groups will be compared using a rate ratio (ratio of negative binomial rates).

Secondary Objectives: 1) Evaluate the impact of a patient-centered discharge instruction tool on health outcomes following hospital discharge. 2) Identify the level of patient and system engagement needed when providing discharge instructions and patient-specific characteristics that might impact the use and effectiveness of discharge instructions.

Secondary Outcome Measures: Self-reported adherence to medications, diet and activity restrictions, and scheduled visits with primary care physician and/or specialist at 30 days following discharge, and a composite of unscheduled visits to primary care physician, emergency room, readmission to hospital or death at 30 days and 3 months following discharge. Proportion of patients who responded "Yes", or "Quite a Bit" or "Completely", to 4 out of the 6 prespecified questions on patient experience of transitions of care, 72 hours following discharge from hospital as a measure of patient experience of their transition of care (original primary outcome, re-specified as secondary outcome based on DMC recommendation).

Study Design: The study will use a mixed methods approach with a randomized controlled trial (RCT) and qualitative study.

Inclusion Criteria: All patients (>=18 years) admitted to inpatient units at University Health Network (UHN) (and other participating hospitals in Ontario) with a primary diagnosis of chronic obstructive pulmonary disease, pneumonia, stroke, congestive heart failure, post hip and knee replacement will be recruited for randomization to receive the PODS versus standard of discharge care. These diseases were chosen to align with the Ministry of Health and Long Term Care (MOHLTC) quality based procedures.

Exclusion Criteria: Patients who are being discharged to another facility rather than home, who have a prognosis of less than 3 months, who do not have a telephone for post-discharge follow-up or with cognitive impairment or significant language barrier for whom a family member or professional interpreter is not available will be excluded from the study.

Intervention: The patient-oriented discharge summary (PODS) is a discharge instruction tool co-created with patients which provides a written template for providers to engage patients and caregivers when reviewing discharge instructions on medications, activity and diet restrictions, follow-up appointments or outstanding investigations and worrisome symptoms warranting emergency care (Appendix A). The PODS also uses plain and simple wording, large fonts, pictograms, and includes white space for patients to take notes and provides the option for translation of major headings into the most common spoken languages. As this will be a pragmatic design, we may make modifications to the process involved in completing the PODS, such as using pre-filled disease-specific information, if system processes and providers involved deem it more usable and feasible.

Sample Size: We estimate that we will require at minimum 199 and at maximum 388 patients in each study arm if we want to detect a 10% minimum improvement in patient experience scores. Currently, we have study centers that would like to participate in Toronto, Ottawa and Thunder Bay.

Accrual Period: Enrollment for this study will begin once ethics approval is obtained and continue until 776 patients have been enrolled (in total across all participating sites).

Study Duration: The study is expected to run between December 1, 2015 and March 31, 2018 (approximately 3 years) following research ethics board (REB) approval. This will allow for a year of study enrollment across participating sites until sample size is achieved as well as 3 months of follow-up for primary and secondary endpoints and a year for data analysis and manuscript preparation.

Data Monitoring Committee (DMC): A DMC was established on May 4, 2018, due to challenges in recruitment and widespread implementation of the intervention across multiple hospitals in Ontario resulting in a change in the standard of discharge care in the trial's setting. In view of the challenges in recruiting future patients, resource constraints, and statistical considerations, the DMC recommended that recruitment be stopped prematurely and that the analytical approach for the primary outcome be changed, analyzing the data as count data rather than dichotomized data. Study recruitment was stopped at the end of August 2018, after a total of 526 participants had been randomized, with final follow up of participants in December 2018 (see the Document Section for full details).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* Able and willing to provide informed consent or have a substitute decision maker that can provide consent and agree to answer follow up as the patient's caregiver
* Admitted to hospital with either congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), Stroke, Pneumonia, Hip Fracture, Knee Replacement or Hip Replacement
* Being discharged home or to a retirement home
* Have a Telephone for post-discharge follow-up

Exclusion Criteria:

* Patients who have already received the PODS in the past
* Being discharged to nursing home, long-term care facility, rehabilitation or other hospital.
* Unable to communicate due to cognitive impairment or language barrier with no caregiver or interpreter available
* Palliative patient with life expectancy <= 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Patient experience of transition of care | 72 hours post-discharge
  Count of negative responses to 6 questions, with first 5 from CIHI CPES-IC: 1.During this hospital stay, did doctors, nurses or other hospital staff talk with you about whether you would have the help you needed when you left the hospital? 2.During this hospital stay, did you get information in writing about what symptoms or health problems to look out for after you left the hospital? 3.Before you left the hospital, did you have a clear understanding about all of your prescribed medications, including those you were taking before your hospital stay? 4.Did you receive enough information from hospital staff about what to do if you were worried about your condition or treatment after you left the hospital? 5.When you left the hospital, did you have a better understanding of your condition than when you entered? 6.When you left the hospital, did you have a clear understanding about your follow-up appointments and investigations? Analysis change via DMC recommendation.

SECONDARY OUTCOMES:
medication adherence | 30 and 90 days
  self-reported adherence to all medications
diet adherence | 30 and 90 days
  self-reported adherence to diet restrictions
activity adherence | 30 and 90 days
  self-reported adherence to activity restrictions
appointment adherence | 30 and 90 days
  self-reported adherence to scheduled appointments
unscheduled utilization | 30 and 90 days
  a binary composite outcome of any unscheduled visits to primary care physician, emergency room, readmission to hospital or death
Patient experience measure [original primary outcome measure] | 72 hours post-discharge
  Proportion of patients who responded "Yes", or "Quite a Bit" or "Completely", to 4 out of the 6 prespecified questions on patient experience of transitions of care, 72 hours following discharge from hospital as a measure of patient experience of their transition of care (original primary outcome, re-specified as secondary outcome based on DMC recommendation).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Okrainec, MD, Principal Investigator — UHN; Howard B Abrams, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada